CLINICAL TRIAL: NCT01765816
Title: Generation 100: How Exercise Affects Mortality and Morbidity in the Elderly: A Randomized Control Study
Brief Title: Generation 100: Blood Volume and Cardiac Function in Healthy Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: Gen-100-sub1
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Ageing
Keywords: Exercise; Elderly; Blood volume; Hemoglobin
MeSH Terms: conditions — Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high intensity interval training (Experimental): one interval training session with 1 x 4 and 4 x 4 minutes interval training at 90-95% of peak heart rate
  Interventions: Behavioral: high intensity interval training; Behavioral: moderate intensity training
- moderate intensity training (Active Comparator): 45 minutes of moderate continuous training at 75% of maximal heart rate
  Interventions: Behavioral: high intensity interval training; Behavioral: moderate intensity training

INTERVENTIONS:
Behavioral: high intensity interval training
Behavioral: moderate intensity training

SUMMARY:
Hypothesis: Exercise will reduce morbidity and mortality rates in an elderly population. The extent of reduction will be intensity dependent.

As part of the "Generation 100" study, this sub-study project will investigate the effect of exercise on blood volume, cardiopulmonary health and heart function in healthy aging. Objective is to determine the acute effect of one endurance training session on blood volume in healthy elderly. The working hypothesis is that one interval training session increases total blood volume by 10% in healthy elderly, and that there will be no change after moderate continuous training.

ELIGIBILITY:
Inclusion Criteria:

* ability to walk at least 1km,
* born in 1938,1939,1940,1941 or 1942
* Sufficiently good health to be able to take part in the study, as determined by the researchers

Exclusion Criteria:

* Illness or disability that precludes exercise or hinders completion of the study
* Uncontrolled hypertension
* Symptomatic valve disease, hyper tropic cardio-myopathy or unstable angina
* Active cancer
* Test results indicating that study participation is unsafe
* Inclusion in other studies conflicting with participation in this one

Ages: 70 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-08; Primary Completion 2014-02 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
total blood volume | 24 hours
  carbon monoxide-rebreathing spirometry (Bayreuth, Germany)

SECONDARY OUTCOMES:
hemoglobin volume | 24 hours
  carbon monoxide-rebreathing spirometry (Bayreuth, Germany)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Wisløff, Professor, Study Chair — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- See also: Generation 100 web page — http://www.ntnu.edu/cerg/generation100